CLINICAL TRIAL: NCT07190898
Title: The Effectiveness of Core and Functional Strength Exercises in Preventing Low Back and Neck Pain in Healthy Women
Brief Title: The Role of Core and Functional Exercises in Low Back and Neck Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Batman University (Other)
Responsible Party: Principal Investigator, merve yiğit kocamer, lecturer, Batman University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BAU-FTR-MYK-02
Record Dates: First submitted 2025-09-17; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Low Back Pain; Neck Pain; Core Exercises Training; Functional Exercise Training
Keywords: low back pain; neck pain; core exercises training; functional exercise training; healthy women; daily activity
MeSH Terms: conditions — Low Back Pain; Neck Pain

STUDY DESIGN:
Intervention Model Description: 1. Core exercises group
  2. Functional strength exercises group
  3. Education Group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- core exercises group (Active Comparator): The participants performed a total of 18 exercise sessions, three times per week over six weeks. All sessions were supervised by a specialist physiotherapist and lasted approximately 45 minutes. Each session consisted of three parts: warm-up, main exercises, and cool-down. The warm-up included low-intensity mobilization and stretching movements. The main part involved plank, side plank, bridge, quadruped balance, and posture-focused exercises. Each exercise was individualized in terms of repetitions and duration according to the participant's capacity. The program was updated every two weeks by adding a new type of exercise. In the cool-down phase, stretching, breathing techniques, and relaxation exercises were performed.
  Interventions: Other: core exercises
- functional strenght exercises (Active Comparator): The participants performed a total of 18 exercise sessions, three times per week over six weeks. All sessions were supervised by a specialist physiotherapist and lasted approximately 45 minutes. Each session consisted of three parts: warm-up, main exercises, and cool-down. The warm-up included joint mobilization and low-intensity aerobic movements. The main part involved functional movements such as sit-to-stand, lunge, squat, step-up, and balance-focused exercises. The difficulty level of the exercises was adjusted according to the participant's capacity, and new exercises were added to the program every two weeks. In the cool-down phase, stretching, breathing techniques, and relaxation exercises were performed.
  Interventions: Other: functional strength exercises
- education group (Active Comparator): On the first day of the study, participants received an educational session on lifestyle modifications related to healthy living and women's health. During the session, information was provided on proper posture, ergonomic movements, the importance of posture in daily life, and pain management. After the completion of the study, the Education Group was directed to either the Core and Postural Stabilization Exercise Program or the Functional Strength Exercise Program, according to their preference.
  Interventions: Other: education group

INTERVENTIONS:
Other: core exercises — The participants performed core exercises three times per week for a total of six weeks
  Arms: core exercises group
Other: functional strength exercises — The participants performed functional strength exercises three times per week for a total of six weeks.
  Arms: functional strenght exercises
Other: education group — During the educational session, participants were provided with information on proper posture, ergonomic movements, the importance of posture in daily life, and pain management.
  Arms: education group

SUMMARY:
Low back and neck pain are common health problems that can negatively affect daily life activities in healthy women. A significant proportion of adults worldwide experience low back or neck pain at some point in their lives, leading to loss of physical function, reduced work capacity, and decreased quality of life. Women who work at desk-based jobs are particularly prone to such pain due to prolonged sitting, computer use, and non-ergonomic postures. Poor posture habits, weak core muscles, and low postural awareness are among the main causes of low back and neck pain. Strengthening the core muscles, enhancing spinal and pelvic stability, improving muscular endurance, and increasing postural awareness are effective methods to reduce the risk of low back and neck pain. Functional strength exercises support safe and effective movement in daily life activities by improving muscle strength, endurance, and coordination. These exercises are important not only for treating existing pain but also as part of preventive health strategies. Preventive exercise programs can reduce the risk of pain and functional loss in healthy individuals, thereby improving long-term quality of life. Although various exercise approaches have been examined in the literature for the prevention of low back and neck pain, studies comparing core and postural stabilization exercises with functional strength exercises in healthy women are limited. This gap does not provide physiotherapists and health professionals with clear evidence on which exercise approach is more effective. This study aims to compare the effects of core and postural stabilization exercises versus functional strength exercises on the risk of low back and neck pain during daily activities in healthy women. The findings of this study are expected to guide the design and implementation of preventive exercise programs for healthy women.

DETAILED DESCRIPTION:
The aim of this study is to compare the effects of core and postural stabilization exercises and functional strength exercises onthe risk of low back and neck pain during daily activities in healthy women. The study was designed as a single-blind randomized controlled trial. Healthy women aged 20-40 years were included in the study.A total of 45 participants, with 15 in each group, took part in the study. Randomization was performed using a computer-generated randomization list. Individuals who agreed to participate were first evaluated for eligibility according to the study's inclusion and exclusion criteria. Eligible participants were then randomly assigned to one of three groups with an equal allocation ratio (1:1:1).One day after the initial assessment, participants received an educational session on lifestyle modifications related to healthy living and women's health. The Core and Postural Stabilization Exercise Group and the Functional Strength Exercise Group performed a total of 18 exercise sessions, three times per week over six weeks. The Education Group, on the other hand, was directed to either the Core and Postural Stabilization or the Functional Strength program according to their preference after the completion of the study.Participants will be evaluated twice: at the beginning of the study and at the end of the 6-week treatment.

ELIGIBILITY:
Inclusion Criteria:

* Absence of any chronic musculoskeletal, neurological, or cardiovascular disorders,
* Not engaging in regular exercise or performing physical activity less than twice a week,
* Presence of low back or neck pain not attributable to pathology during daily activities,
* No history of major orthopedic surgery within the last six months.

Exclusion Criteria:

* Individuals with severe orthopedic, neurological, or cardiovascular diseases,
* Those who have undergone surgical interventions involving the lumbar or cervical regions within the past six months,
* Individuals who regularly participate in physiotherapy or structured exercise programs.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 45 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Nordic Musculoskeletal Questionnaire (NMQ) | 6 week
  An internationally recognized questionnaire used to assess musculoskeletal symptoms. It specifically asks about pain, discomfort, and limited movement in areas such as the back, neck, and shoulders. The questionnaire divides the body into nine anatomical regions and asks whether pain, discomfort, or limited movement has been experienced in the last 12 months and the last 7 days. A higher score indicates greater prevalence and frequency of pain.
Visual Analog Scale (VAS) | 6 week
  This is a simple and reliable self-report scale used to measure pain intensity. The participant is usually shown a 10 cm long line; one end of the line represents "no pain" (0), and the other end represents "unbearable pain" (10). The participant marks a point on the line according to the intensity of pain they are currently experiencing. Pain intensity is numerically determined by measuring the position of the mark on the line.
Oswestry Disability Index (ODI) | 6 week
  This 10-section scale covers topics such as pain intensity, personal care, lifting, walking, sitting, standing, sleeping, social life, travel, and sexual life. Each section is scored from 0 to 5. A higher total score indicates a greater degree of functional disability due to low back pain. Results from the scale are expressed as percentages, with 0-20% representing minimal disability, 21-40% representing moderate disability, 41-60% representing severe disability, 61-80% representing severe disability, and 81-100% representing complete dependency.
Neck Disability Index (NDI) | 6 week
  This is a valid and reliable scale widely used in clinical and research settings that measures the impact of neck pain on individuals' activities of daily living. This 10-section scale covers topics such as pain intensity, personal care, lifting, reading, headache, concentration, working, driving, sleep, and recreational activities. Each section is scored from 0 to 5. As the total score increases, the functional disability associated with neck pain increases. The resulting score is expressed as a percentage, with 0-20% representing minimal disability, 21-40% representing moderate disability, 41-60% representing severe disability, 61-80% representing severe disability, and 81-100% representing complete dependency.

SECONDARY OUTCOMES:
Functional Movement Screen (FMS) | 6 week
  The FMS is a valid and reliable assessment tool that examines an individual's basic movement patterns and is used to determine movement quality and potential injury risk. It consists of seven different tests: deep squat, hurdle step, in-line lunge, shoulder mobility, active straight leg raise, trunk stability push-up, and rotary stability. Each movement is scored from 0 to 3, with a total score ranging from 0 to 21. Lower scores indicate functional movement limitations and a higher risk of injury, while higher scores indicate better movement quality and postural control.
Plank and Side Plank Tests | 6 week
  The plank test measures how long an individual can maintain a correct plank position on their forearms and toes, and this time is recorded in seconds. The side plank test measures the time an individual can maintain a side plank position to assess the lateral core muscles. Both tests provide information about the isometric endurance of the core muscles. The longer the duration, the better the core endurance.
Sit-to-Stand Test | 6 week
  In this test, the individual is asked to sit down and stand up from a chair as many times as possible within a specific time period (e.g., 30 seconds), or the time taken to complete five repetitions of the sit-to-stand movement is recorded. The resulting value provides information about lower extremity strength, functional independence, and mobility. A shorter time or a greater number of repetitions indicates better lower extremity strength and functional capacity.

CONTACTS AND LOCATIONS:
Overall Officials: merve yiğit kocamer, lecturer, Principal Investigator — Batman University
Locations (2):
- Turkey (Türkiye) (2):
  - Batman University, Batman, Batman
  - Batman Center, Batman, Gültepe

IPD SHARING:
Plan to Share IPD: No